CLINICAL TRIAL: NCT00806637
Title: Vessel Sealing System Uvulopalatoplasty vs Uvulopalatal Flap: a Randomized, Control Study of Efficacy and Adverse Effects
Brief Title: Vessel Sealing System Uvulopalatoplasty Versus Uvulopalatal Flap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chulalongkorn University (Other)
Responsible Party: Prakobkiat Hirunwiwatkul, Department of Otolaryngology, Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENTCU_pkk2008_02
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-10

CONDITIONS: Snoring; Obstructive Sleep Apnea
Keywords: Vessel sealing system; uvulopalatoplasty; UPPP; uvulopalatal flap; bleeding; operative time; adverse effects
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Vessel sealing system uvulopalatoplasty (VSSU) is a new technique for uvulopalatoplasty using a special biclamp forceps for better hemostasis control. Vessel sealing system (VSS) is a bipolar vascular sealing system, with integrated active feedback control. The tissue is grasped and compressed by the handpiece. After the instrument is removed, the seal is visible as a semitransparent window, which can safely be divided. Uvular tip is grasped with an Allis clamp and retracted back toward the soft palate. Excision of the uvula and the redundant part of soft palate is performed by the VSS handpiece. VSS is also used for hemostasis.
  Interventions: Procedure: Vessel sealing system uvulopalatoplasty (VSSU)
- 2 (Active Comparator): Uvulopalatal flap (UPF) is a standard uvulopalatoplasty technique. Uvulopalatal flap is usually performed as described originally by Powell et al. The soft palate was injected with 5 to 10 milliliters of 1% lidocaine with epinephrine solution. The mucosa, submucosa with glands, and fat on the lingual surface of the uvula and soft palate were removed with a scalpel. Bleeding was controlled with bipolar electrocoagulation. The uvular tip was amputated, and reflected back toward the soft palate, and fixated into its new position with multiple sutures of 3-0 chromic catgut.
  Interventions: Procedure: Uvulopalatal flap (UPF)

INTERVENTIONS:
Procedure: Vessel sealing system uvulopalatoplasty (VSSU) — Vessel sealing system uvulopalatoplasty (VSSU) is a new technique for uvulopalatoplasty using a special biclamp forceps for better hemostasis control. Vessel sealing system (VSS) is a bipolar vascular sealing system, with integrated active feedback control. The tissue is grasped and compressed by the handpiece. After the instrument is removed, the seal is visible as a semitransparent window, which can safely be divided. Uvular tip is grasped with an Allis clamp and retracted back toward the soft palate. Excision of the uvula and the redundant part of soft palate is performed by the VSS handpiece. VSS is also used for hemostasis.
  Other Names: ligasure vessel sealing system
  Arms: 1
Procedure: Uvulopalatal flap (UPF) — Uvulopalatal flap (UPF) is a standard uvulopalatoplasty technique. Uvulopalatal flap is usually performed as described originally by Powell et al. The soft palate was injected with 5 to 10 milliliters of 1% lidocaine with epinephrine solution. The mucosa, submucosa with glands, and fat on the lingual surface of the uvula and soft palate were removed with a scalpel. Bleeding was controlled with bipolar electrocoagulation. The uvular tip was amputated, and reflected back toward the soft palate, and fixated into its new position with multiple sutures of 3-0 chromic catgut.
  Other Names: uvulopalatoplasty
  Arms: 2

SUMMARY:
The purpose of this study is to compare vessel sealing system uvulopalatoplasty (VSSU) to the traditional uvulopalatal flap (UPF) in the treatment of sleep-disordered breathing with special regard to intraoperative bleeding, operative time, postoperative pain, postoperative hemorrhage and other adverse effects.

DETAILED DESCRIPTION:
Uvulopalatopharyngoplasty is one of the common procedures performed by otolaryngologists to treat sleep-disordered breathing patients who have retropalatal obstruction. Intraoperative bleeding is a significant problem which requires hemostasis and causes prolonged operative time. Several different techniques are used to perform this operation, including cold knife, monopolar cautery, coblation, and radiofrequency. Efficacy in hemostasis and tissue trauma from different operative techniques may result in different operative time and different degrees of morbidity including intraoperative blood loss, postoperative pain, postoperative hemorrhage, and velopharyngeal insufficiency (VPI). The vessel sealing system has been widely used in head and neck surgery because of its effectiveness and safety. It was also found quite effective and safe in tonsillectomy procedures, providing excellent hemostasis and minimal tissue trauma.

ELIGIBILITY:
Inclusion Criteria:

* Patient planned for uvulopalatoplasty for indications of snoring or obstructive sleep apnea
* Written informed consent form is given from patient

Exclusion Criteria:

* Pregnancy
* History of bleeding disorders
* Patient unable to understand evaluation method
* Patient unable to be contacted via telephone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | within the first 1 hour after surgery starting time

SECONDARY OUTCOMES:
operative time | within the first 1 hour after surgery starting time
postoperative pain | within the first 14 days after surgery
postoperative bleeding | within the first 14 days after surgery
postoperative velopharyngeal insufficiency | within the first 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Prakobkiat Hirunwiwatkul, M.D., Principal Investigator — Department of Otolaryngology, Faculty of Medicine, Chulalongkorn University
Locations (1):
- Department of Otolaryngology, Faculty of Medicine, Chulalongkorn University, Patumwan, Bangkok, Thailand

REFERENCES:
- [Result] Lachanas VA, Hajiioannou JK, Karatzias GT, Filios D, Koutsias S, Mourgelas C. Comparison of LigaSure vessel sealing system, harmonic scalpel, and cold knife tonsillectomy. Otolaryngol Head Neck Surg. 2007 Sep;137(3):385-9. doi: 10.1016/j.otohns.2007.05.012. PMID 17765762
- [Result] Powell N, Riley R, Guilleminault C, Troell R. A reversible uvulopalatal flap for snoring and sleep apnea syndrome. Sleep. 1996 Sep;19(7):593-9. doi: 10.1093/sleep/19.7.593. PMID 8899940
- [Result] Prokopakis EP, Lachanas VA, Helidonis ES, Velegrakis GA. The use of the Ligasure Vessel Sealing System in parotid gland surgery. Otolaryngol Head Neck Surg. 2005 Nov;133(5):725-8. doi: 10.1016/j.otohns.2005.06.030. PMID 16274800
- [Result] Bassiouny A, El Salamawy A, Abd El-Tawab M, Atef A. Bipolar radiofrequency treatment for snoring with mild to moderate sleep apnea: a comparative study between the radiofrequency assisted uvulopalatoplasty technique and the channeling technique. Eur Arch Otorhinolaryngol. 2007 Jun;264(6):659-67. doi: 10.1007/s00405-007-0244-x. Epub 2007 Feb 9. PMID 17294208